CLINICAL TRIAL: NCT00046566
Title: Clinical Trial of Dietary Protein on Blood Pressure
Brief Title: Clinical Trial of Dietary Protein and Blood Pressure
Acronym: ProBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Professor and Chair, Tulane University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 145; R01HL068057 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases

STUDY DESIGN:
Intervention Model Description: The trial participants were assigned to take 40 g/d soy protein, milk protein, or carbohydrate supplementation each for 8 weeks in a random order. A 3-week washout period was implemented between the interventions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization assignment list was generated by a computer program that could only be accessed by the study data coordinator. Apart from the data coordinator, all research personnel, including study coordinators and BP technicians, and the study participants were unaware of treatment assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Soy protein-milk protein-carbohydrate (Active Comparator): Participants received 40 grams of soy protein daily for 8 weeks, 40 grams of milk protein daily for 8 weeks, and 40 grams of carbohydrate daily for 8 weeks.
  Interventions: Dietary Supplement: Soy protein-milk protein-carbohydrate
- Milk protein-carbohydrate-soy protein (Experimental): Participants received 40 grams of milk protein daily for 8 weeks, 40 grams of carbohydrate daily for 8 weeks, and 40 grams of soy protein daily for 8 weeks.
  Interventions: Dietary Supplement: Milk protein-carbohydrate-soy protein
- Carbohydrate-soy protein-milk protein (Placebo Comparator): Participants received 40 grams of complex carbohydrate daily for 8 weeks, 40 grams of soy protein daily for 8 weeks, and 40 grams of milk protein daily for 8 weeks.
  Interventions: Behavioral: Carbohydrate-soy protein-milk protein

INTERVENTIONS:
Dietary Supplement: Soy protein-milk protein-carbohydrate — 40 grams of soy protein per day for 8 weeks, 40 grams of milk protein per day for 8 weeks, and 40 grams of carbohydrate per day for 8 weeks
  Arms: Soy protein-milk protein-carbohydrate
Dietary Supplement: Milk protein-carbohydrate-soy protein — 40 grams of milk protein per day for 8 weeks, 40 grams of carbohydrate per day for 8 weeks, 40 grams of soy protein per day for 8 weeks.
  Arms: Milk protein-carbohydrate-soy protein
Behavioral: Carbohydrate-soy protein-milk protein — 40 grams of carbohydrate per day for 8 weeks, 40 grams of soy protein per day for 8 weeks, 40 grams of milk protein per day for 8 weeks,
  Arms: Carbohydrate-soy protein-milk protein

SUMMARY:
The purpose of this study is to examine the effect of dietary protein supplements on high blood pressure (BP).

DETAILED DESCRIPTION:
BACKGROUND:

At least 50 million adult Americans have high BP, which is one of the most important modifiable risk factors for coronary heart disease, stroke, and end-stage kidney disease. Nutrient intake has been related to the development of high BP, and nutritional modifications have become an important approach for the treatment and prevention of high BP. While the effect of sodium, potassium, and alcohol on BP has been studied extensively, the effect of dietary macronutrients, such as protein, has not been as well studied. Results from this study may provide justification for recommending protein supplements for the prevention and treatment of high BP in the general population.

DESIGN NARRATIVE:

The study will enroll 280 healthy participants with BP levels higher than optimal or with stage-1 hypertension (systolic BP of 120-159 mm Hg and diastolic BP of 80-95 mm HG). Participants will be recruited by a mass mailing and a worksite/community-based BP screening in New Orleans, Louisiana, and Jackson, Mississippi. Following a two-week screening period, eligible participants will receive either 40 grams of soy protein, 40 grams of milk protein, or 40 grams of complex carbohydrates (control) daily for eight weeks. Following those eight weeks, participants will not receive any supplements for three weeks. Participants will then repeat the process with the other two supplements. The primary outcome will be difference in BP during the soy protein supplementation, milk protein supplementation, and placebo control phases. In addition, changes in serum lipids; waist and hip circumference; and fasting plasma insulin, glucose, leptin, and homocysteine will be monitored and examined in terms of impact on BP level.

ELIGIBILITY:
Inclusion Criteria:

* Systolic BP of 120 to 159 mm Hg and diastolic BP of 80 to 95 mm Hg (average of 6 measurements at 2 screening visits)
* Willing to participate in all aspects of the study

Exclusion Criteria:

* Consumption of dietary protein greater than or equal to 1.63 grams/kg per day, as determined by two 24-hour dietary recalls
* Stage-2 or higher severe hypertension (systolic BP greater than or equal to 160 mm Hg and/or diastolic BP greater than or equal to 95 mm Hg)
* Use of antihypertensive medications or medications that affect BP
* History of clinical heart disease (e.g., angina/heart attack, coronary revascularization, heart failure, stroke/transient ischemic attack, peripheral arterial disease)
* Kidney disease (serum creatinine level greater than or equal to 1.7 mg/dL for men and greater than or equal to 1.5 mg/dL for women)
* Current hypercholesterolemia (fasting serum total cholesterol greater than or equal to 240 mg/dL) or use of cholesterol-lowering medications
* Current diabetes (fasting serum glucose greater than or equal to 126 mg/dL) or use of insulin or oral hypoglycemic agents
* Severe obesity (body mass index greater than or equal to 40 kg/m²)
* Current use of prescription weight loss medications, underwent weight loss surgery, and/or experienced weight loss greater than 15 pounds within the 6 months prior to study entry
* Cancer (except non-melanoma skin cancer) that required treatment during the year prior to study entry
* Consumption of more than 14 alcoholic beverages per week
* Current participation in another medical study
* Consumption of milk or soy protein greater than or equal to the 90th percentile of intake in the U.S. general population
* Has another member of the household participating in the study
* Study employees or living with study employees
* Allergy or intolerance to soy protein or milk protein products
* Allergy to aspartame
* Plans to move out of the study area (greater than or equal to 50 miles from the study site) and has difficulty coming to the study site
* Inability or unwillingness to cooperate during the screening visits
* Poor compliance during the screening period (intake of less than 85% of supplements)
* Pregnant or plans to become pregnant during the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2002-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, Study Chair — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Rebholz CM, Reynolds K, Wofford MR, Chen J, Kelly TN, Mei H, Whelton PK, He J. Effect of soybean protein on novel cardiovascular disease risk factors: a randomized controlled trial. Eur J Clin Nutr. 2013 Jan;67(1):58-63. doi: 10.1038/ejcn.2012.186. Epub 2012 Nov 28. PMID 23187956
- [Result] He J, Wofford MR, Reynolds K, Chen J, Chen CS, Myers L, Minor DL, Elmer PJ, Jones DW, Whelton PK. Effect of dietary protein supplementation on blood pressure: a randomized, controlled trial. Circulation. 2011 Aug 2;124(5):589-95. doi: 10.1161/CIRCULATIONAHA.110.009159. Epub 2011 Jul 18. PMID 21768541
- [Result] Wofford MR, Rebholz CM, Reynolds K, Chen J, Chen CS, Myers L, Xu J, Jones DW, Whelton PK, He J. Effect of soy and milk protein supplementation on serum lipid levels: a randomized controlled trial. Eur J Clin Nutr. 2012 Apr;66(4):419-25. doi: 10.1038/ejcn.2011.168. Epub 2011 Sep 28. PMID 21952693

RESULTS

PARTICIPANT FLOW:
Groups:
- Soy Protein-milk Protein-carbohydrate Group: 117 participants assigned to soy protein-milk protein-carbohydrate group. They received 40 g/d soy protein for 8 weeks, then 40 g/d milk protein for 8 weeks, and finally 40 g/d carbohydrate for 8 weeks.
- Milk Protein-carbohydrate-soy Protein Group: 117 participants assigned to milk protein-carbohydrate-soy protein group. They received 40 g/d milk protein for 8 weeks, then 40 g/d carbohydrate for 8 weeks, and finally 40 g/d soy protein for 8 weeks.
- Carbohydrate-soy Protein-milk Protein Group: 118 participants assigned to carbohydrate-soy protein-milk protein group. They received 40 g/d carbohydrate for 8 weeks, then 40 g/d soy protein for 8 weeks, and finally 40 g/d milk protein for 8 weeks.
Period: Intervention 1 (8 Weeks)
Arm/Group | Soy Protein-milk Protein-carbohydrate Group | Milk Protein-carbohydrate-soy Protein Group | Carbohydrate-soy Protein-milk Protein Group
Started | 117 (Soy protein 8 weeks) | 117 (Milk protein 8 weeks) | 118 (Carbohydrate 8 weeks)
Completed | 101 | 104 | 101
Not Completed | 16 | 13 | 17
Period: Intervention 2 (8 Weeks)
Arm/Group | Soy Protein-milk Protein-carbohydrate Group | Milk Protein-carbohydrate-soy Protein Group | Carbohydrate-soy Protein-milk Protein Group
Started | 101 (Milk protein 8 weeks) | 104 (Carbohydrate 8 weeks) | 101 (Soy protein 8 weeks)
Completed | 93 | 92 | 88
Not Completed | 8 | 12 | 13
Period: Intervention 3 (8 Weeks)
Arm/Group | Soy Protein-milk Protein-carbohydrate Group | Milk Protein-carbohydrate-soy Protein Group | Carbohydrate-soy Protein-milk Protein Group
Started | 93 | 92 | 88
Completed | 93 | 92 | 88
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Soy Protein-milk-protein-carbohydrate: Soy protein-milk-protein-carbohydrate group
- Milk Protein-carbohydrate-soy Protein: Milk protein-carbohydrate-soy protein group
- Carbohydrate-soy Protein-milk Protein: Carbohydrate-soy protein-milk protein group
- Total: Total of all reporting groups
Arm/Group | Soy Protein-milk-protein-carbohydrate | Milk Protein-carbohydrate-soy Protein | Carbohydrate-soy Protein-milk Protein | Total
Number analyzed (Participants) | 117 | 117 | 118 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.5) | 46.7 (10.7) | 48.1 (8.7) | 47.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 68 | 205
  Male | 48 | 49 | 50 | 147
Region of Enrollment [Number; unit: participants]
  United States | 117 | 117 | 118 | 352

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Systolic Blood Pressure at 8 Weeks
Description: The change of systolic blood pressure was calculated as the mean of 6 blood pressure values from two 8-week visits minus the mean of 6 values from two baseline visits within each intervention phase. At each visit, 3 BP values were measured with a Hawksley random-zero sphygmomanometer by trained and certified observers who were masked to group assignment. BP readings were taken from the right arm with appropriately sized cuffs after the participant had been seated quietly for 5 minutes. The participant was instructed not to eat, smoke, drink alcohol, or exercise for at least 30 minutes before their BP measurements.
Time Frame: Every 8 weeks
Population: participants took soy protein during three phases
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Soy Protein Supplementation: Cross-over analysis of soy protein supplementation
- Milk Protein Supplementation; Carbohydrate Supplementation: Cross-over analysis of milk protein supplementation
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
Number analyzed (Participants) | 284 | 286 | 287
mmHg | -1.5 [-2.4 to -0.6] | -1.8 [-2.7 to -1.0] | 0.5 [-0.4 to 1.3]

2. Secondary Outcome: Change From Baseline in Serum LDL-cholesterol at 8 Weeks
Description: Change in serum LDL-cholesterol was calculated as LDL-cholesterol at 8 weeks minus LDL-cholesterol at baseline. Over-night fasting serum LDL-cholesterol was measured with an enzymatic method.
Time Frame: Every 8 weeks
Population: Participants took soy protein for 8 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Carbohydrate Supplementation: Cross-over analysis carbohydrate supplementation
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
Number analyzed (Participants) | 284 | 286 | 287
mg/dL | -3.97 [-7.63 to -0.31] | -2.56 [-5.40 to 0.28] | -1.41 [-4.24 to 1.42]

3. Secondary Outcome: Body Weight at 8 Weeks
Description: Body weight was measured by trained staff using a standard protocol at week 8.
Time Frame: Every 8 weeks
Population: Participants took supplementation for 8 weeks
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
Number analyzed (Participants) | 310 | 306 | 315
kg | 86.2 [84.4 to 88.0] | 86.6 [84.9 to 88.4] | 86.7 [84.9 to 88.5]

ADVERSE EVENTS:
Time Frame: From date of randomization until the date of study withdrawal or completion, whichever came first, assessed every 8 weeks, up to 24 weeks.
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
All-Cause Mortality (participants affected / at risk) | 0/284 | 0/286 | 0/287
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/286 | 0/287
Other Adverse Events (participants affected / at risk) | 0/284 | 0/286 | 0/287

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes